CLINICAL TRIAL: NCT04149938
Title: Phase 1, Randomized Comparative Pharmacokinetic Study of Lidocaine Patch 1.8% (ZTlido™) and Lidocaine Patch 5% (Lidoderm®) in Healthy Subjects
Brief Title: Comparative Pharmacokinetic Study of Lidocaine Patch 1.8% (ZTlido™) and Lidocaine Patch 5% (Lidoderm®) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SCI-LIDO-PK-002A
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine; Lidoderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lidocaine Patch (Sequence AB) (Experimental): Subjects received all study treatments: ZTlido and Lidoderm. On Day 1 (Period 1), three ZTlido lidocaine topical systems were applied to the skin on the back for 12 hours. On Day 8 (Period 2), three Lidoderm lidocaine patches were applied to the skin on the back for 12 hours.
  Interventions: Drug: Lidocaine topical system 1.8%; Drug: Lidocaine patch 5%
- Lidocaine Patch (Sequence BA) (Experimental): Subjects received all study treatments: ZTlido and Lidoderm. On Day 1 (Period 1), three Lidoderm lidocaine patches were applied to the skin on the back for 12 hours. On Day 8 (Period 2), three ZTlido lidocaine topical systems were applied to the skin on the back for 12 hours.
  Interventions: Drug: Lidocaine topical system 1.8%; Drug: Lidocaine patch 5%

INTERVENTIONS:
Drug: Lidocaine topical system 1.8%
  Other Names: Lidocaine patch 1.8%; ZTlido
Drug: Lidocaine patch 5%
  Other Names: Lidoderm

SUMMARY:
The purpose of this study is to characterize the comparative single-dose pharmacokinetics (bioequivalence) of lidocaine patch 1.8% (investigational product) versus Lidoderm® (lidocaine patch 5%,reference product).

ELIGIBILITY:
Key Inclusion Criteria:

* Must be healthy based on medical history, laboratory work, and physical exam
* Be ≥18 and ≤65 years of age
* Females of childbearing potential must not be pregnant and be using an acceptable form of birth control
* Must be free of any systemic or dermatologic disorder

Key Exclusion Criteria:

* Use of prescription medication within 14 days or over-the-counter products within 7 days prior to study medication
* Current use of opioids
* Known hypersensitivity or allergy to any of the components of the product formulations
* Any serious illness in the 4 weeks preceding the beginning of treatment that resulted in missed work or hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of lidocaine | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Peak plasma concentration of lidocaine after application of 3 patches for 12 hours
Area under the Plasma-Concentration Time Curve (AUC) from Time 0 to Time 48 hours | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Area under the plasma concentration versus time curve from 0 to 48 hours of lidocaine in plasma
Area under the Plasma-Concentration Time Curve (AUC) from Time 0 to Time Infinity | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Area under the plasma concentration versus time curve from 0 to infinite time of lidocaine in plamsa
Apparent dose | 0 to 12 hours
  Apparent dose of delivered lidocaine assessed by calculating the quantity of lidocaine in the patch as manufactured minus the quantity recovered from the used patch after 12 hours of wear and adhesive residue remaining on skin and on the product liner and envelope

CONTACTS AND LOCATIONS:
Overall Officials: Phillip LaStella, MD, Principal Investigator — TKL Research, Inc.

REFERENCES:
- [Derived] Gudin J, Argoff C, Fudin J, Greuber E, Vought K, Patel K, Nalamachu S. A Randomized, Open-Label, Bioequivalence Study of Lidocaine Topical System 1.8% and Lidocaine Patch 5% in Healthy Subjects. J Pain Res. 2020 Jun 22;13:1485-1496. doi: 10.2147/JPR.S237934. eCollection 2020. PMID 32606914